CLINICAL TRIAL: NCT00045136
Title: A Multicenter Dosimetry Trial to Evaluate Radiation Absorbed Dose From Holmium-166-DOTMP in Patients With Multiple Myeloma
Brief Title: Chemotherapy, Holmium Ho 166 DOTMP, and Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Poniard Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000256377; PONIARD-0102; NEORX-0102; FHCRC-1704.00
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Melphalan; Peripheral Blood Stem Cell Transplantation; holmium-1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetrakis(methylenephosphonic acid)

INTERVENTIONS:
Drug: melphalan
Procedure: peripheral blood stem cell transplantation
Radiation: holmium Ho 166 DOTMP

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Holmium Ho 166 DOTMP may deliver radiation directly to cancer cells and cause less damage to normal tissue. Combining chemotherapy and holmium Ho 166 DOTMP with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy and holmium Ho 166 DOTMP and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining holmium Ho 166 DOTMP with melphalan and peripheral stem cell transplantation in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the radiation absorbed dose of holmium Ho 166 DOTMP to the kidney in patients with multiple myeloma, based on whole body gamma camera image data for comparison with that obtained using an ICRP mathematical model.
* Determine the average marrow dose of this drug in these patients using gamma camera whole body counts in patients receiving this drug.
* Determine the pharmacokinetics of this drug in these patients.
* Compare marrow dose estimates determined from gamma camera whole-body counts and thyroid uptake probe counts in patients receiving this drug.
* Evaluate intra-patient variability of the uptake of this drug in the bone with repeat tests.
* Determine whether the biodistribution and dosimetry is influenced by administering this drug as a bolus compared to a 15-minute infusion in these patients.
* Compare the reduction in dose rate from the 15-minute infusion vs the bolus injection of this drug to estimate the effect on kidney exposure in these patients.
* Determine the renal transit time for each patient after bolus injection of this drug and assess whether this information improves the dose estimate to kidney with the mathematical model.
* Determine whether there is correlation of renal transit time from technetium Tc 99m-diethylenetriaminepentaacetic acid (DTPA) with holmium Ho 166 DOTMP.
* Determine the adverse events in patients receiving this drug.
* Determine the efficacy of a targeted therapy dose of holmium Ho 166 DOTMP with melphalan followed by autologous peripheral blood stem cell transplantation in these patients.

OUTLINE: This is a multicenter study. Patients are entered into one of two cohorts.

* Cohort A: Patients receive a diagnostic dose of holmium Ho 166 DOTMP IV over 15 minutes on day 1 and then IV bolus on day 8.
* Cohort B: Patients receive a diagnostic dose of holmium Ho 166 DOTMP IV over 15 minutes on days 1 and 8.

After each diagnostic dose, patients in both cohorts also undergo gamma camera imaging of the whole body on days 1 and 8.

Approximately 1-3 weeks later, patients in both cohorts who demonstrate adequate uptake of the first diagnostic dose of holmium Ho 166 DOTMP into the bone marrow then receive therapeutic holmium Ho 166 DOTMP IV over 15 minutes once between days -13 to -10 followed by melphalan IV over 20-30 minutes once between days -10 to -1. Patients undergo autologous peripheral blood stem cell transplantation on day 0.

Patients are followed monthly for 1 year and then every 3 months for 1 year.

PROJECTED ACCRUAL: A minimum of 12 patients (6 per cohort) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma (MM)

  * Patients with a prior diagnosis of monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma are eligible if they progressed and met the criteria for diagnosis of MM
* No non-secretory MM
* No symptomatic MGUS, smoldering MM, or indolent MM
* No solitary bone or extramedullary plasmacytoma
* No immunoglobulin M myeloma
* Prior induction therapy for myeloma required
* Responding, stable, or progressive disease after induction therapy, or relapsed disease
* Candidate for autologous hematopoietic stem cell transplantation
* Prior stem cell mobilization with chemotherapy and growth factors according to institutional procedures

  * Availability of at least 2,000,000 CD34+ cells/kg

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 2 mg/dL
* SGPT no greater than 2 times upper limit of normal
* No clinical evidence of amyloidosis of the liver

Renal

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 45 mL/min
* Renal ultrasound normal
* No clinical evidence of amyloidosis of the kidney
* No urinary obstruction in the renal pelvis, ureter, or bladder outlet by ultrasound

Cardiovascular

* Ejection fraction at least 50% with no evidence of amyloidosis by echocardiogram
* No clinical evidence of amyloidosis of the heart
* No uncontrolled arrhythmia
* No symptomatic cardiac disease

Pulmonary

* FEV1, FVC, and DLCO at least 60%
* No symptomatic pulmonary disease
* No clinical evidence of amyloidosis of the lungs

Other

* No known allergy to vitamin C or bisphosphonates
* No known hypersensitivity to technetium Tc 99m phosphorus radiopharmaceuticals (e.g., technetium Tc 99m-methylene diphosphonate)
* No concurrent illness that would severely limit life expectancy
* No symptoms, physical findings, or radiographic evidence of cord compression
* No clinical evidence of amyloidosis of the autonomic nervous system or gastrointestinal tract
* No prior noncompliance in other studies
* No other malignancy within the past 5 years except treated indolent skin cancers or carcinoma in situ of the cervix
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior stem cell or bone marrow transplantation
* No concurrent maintenance therapy comprising interferon or thalidomide

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics
* No concurrent maintenance therapy comprising dexamethasone

Radiotherapy

* No prior cumulative external-beam radiotherapy (EBRT) to more than 20% of bone marrow
* No prior cumulative EBRT dose of 30 Gy or more to the spinal cord
* No prior radiotherapy to the bladder

Surgery

* See Disease Characteristics

Other

* At least 4 weeks since prior investigational agents for MM
* At least 4 weeks since other prior experimental therapies for any other condition
* No bisphosphonates for at least 4 weeks before study, during study, and for at least 30 days posttransplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Jenkins, Principal Investigator — Poniard Pharmaceuticals
Locations (5):
- United States (5):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of California Davis Cancer Center, Sacramento, California
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington